CLINICAL TRIAL: NCT02582710
Title: Impact of an Optimized Formulation of Omega 3 on the Composition of Atheromatous Plaques in Patients Requiring Carotid Endarterectomy
Acronym: POMEGA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5714
Record Dates: First submitted 2015-09-29; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Carotid Endarterectomy
MeSH Terms: interventions — VASCAZEN

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VASCAZEN (Experimental): Patients treated with Vascazen
  Interventions: Dietary Supplement: VASCAZEN
- Placebo (Placebo Comparator): Patients treated with a placebo
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: VASCAZEN — 6 weeks treatment with an optimized formulation of omega 3 before the carotid endarterectomy
  Arms: VASCAZEN
Dietary Supplement: PLACEBO — 6 weeks treatment with a placebo before the carotid endarterectomy
  Arms: Placebo

SUMMARY:
Determining whether treatment with an optimized formulation of omega 3 for 6 weeks causes a 40% decrease in the average concentration of total microparticles (MPs) in the atheromatous plaque.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 30 and 85 years
* Affiliated to a social security scheme
* Informed consent signed
* Patients to get an endarterectomy carotid stenosis> 70% asymptomatic is
* Women of childbearing potential (negative pregnancy test), effective contraception for the duration of the study

Exclusion Criteria:

* Inability to give informed information about the study (subject in emergencies, difficulty of understanding ...)
* Patient treated by OMACOR®
* Patients on oral anticoagulant (AVK, apixaban, dabigatran, rivaroxaban)
* Daily consumption of fish oil (medical food with fish oil (omega 3))
* Carotid Restenosis
* Pregnancy (positive pregnancy test) and lactation
* Hypersensitivity to fish
* Allergy to fish
* Subject under judicial protection
* Subjects under guardianship or curatorship

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related postive event assessed by the reduction of the concentration of procoagulant microparticles in the atherosclortic plaque | an average of 1 to 6 months after the carotid endarterectomy
  Microparticle concentration measured by captured-based prothrombinase assay

SECONDARY OUTCOMES:
Number of participants with treatment-related modification of the content of the plaque assessed by protein biomarkers of the plaque instability and thrombogenicity, and by the identification of the cell origin of the procoagulant microparticles | an average of 1 to 6 months after the carotid endarterectomy
  Number of patients with treatment-related modifications in the concentration of blood biomarkers of thrombogenicity. Comparisons of plaque and blood biomarkers variations related to the treatment Description field : Cell origin of MPs measured prothrombinase assay after capture on cell lineage specific antibodies. Detection of proteases and biomakers by western blot or activity assays.

CONTACTS AND LOCATIONS:
Locations (1):
- Nouvel Hopital Civil, Strasbourg, France